CLINICAL TRIAL: NCT06876350
Title: Patient Satisfaction for Post-Operative Carpometacarpal Arthroplasty: Wood Casting Versus Thermoplastic Splint
Brief Title: Woodcasting Versus Thermoplast Splint in CMC Arthroplasty
Acronym: Woodcast
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Orthopaedic Research and Education (Other)
Responsible Party: Principal Investigator, Michael C. Doarn, Principal Investigator, Foundation for Orthopaedic Research and Education
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Study007574
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Carpometacarpal (CMC) Joint Arthritis
Keywords: Randomized; Hand and Upper Extremity
MeSH Terms: conditions — Capillary Malformations, Congenital, 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Woodcasting Splint (Experimental): Woodcasting is an already FDA approved on the market product that is not used a lot so for the purpose of the study we would like to show superior outcomes.
  Interventions: Other: Woodcasting Splint
- Thermoplastic Splint (Active Comparator): Thermoplastic splints is an FDA approved on the market orthrosis that is used by Occupational Therapists which is standard of care for patients that undergo CMC arthroplasty.
  Interventions: Other: Control (Standard treatment)

INTERVENTIONS:
Other: Woodcasting Splint — This is the experimental group so we could see the outcomes and preference for patients using surveys and compliance scores
  Arms: Woodcasting Splint
Other: Control (Standard treatment) — Thermoplastic splints are standard of care treatment for patients after CMC arthroplasty. We will use the data from this group as the comparator to the experimental group.
  Arms: Thermoplastic Splint

SUMMARY:
This study is a prospective, randomized, nonblinded trial to evaluate patient preference in splints after having a carpometacarpal arthroplasty.

DETAILED DESCRIPTION:
Patients undergoing carpometacarpal arthroplasty will be randomized into the woodcast or thermoplast splint after their surgery to see which is preferred using compliance and surveys.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 years old.
* Intact Medical Decision Making
* Eligible for Surgical Intervention
* Willing to comply with all aspects of the treatment and evaluation schedule over 6 weeks

Exclusion Criteria:

* Pregnant Women
* Deemed Unsuitable by Principal Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction Score | 6 Weeks
  The satisfaction survey consists of three questions totaling 15. The minimum value is a 1, while the maximum value is 15. A higher score indicating highest satisfaction.

SECONDARY OUTCOMES:
Waste | 2 Weeks
  Each splint group creates waste for the fabrication and molding for each patient which will be recorded by the clinical research coordinator and weighed out.
Splint Satisfaction | 6 Weeks
  Patient will have three questions totaling 15 with the higher score indicating highest satisfaction.
Splint Issues | 6 Weeks
  A single question will be filled out by patients on a scale of 1-5 with a score of 5 indicating a lot of issues with their splint.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Doarn, MD, Principal Investigator — Florida Orthopaedic Institute
Locations (1):
- Florida Orthopaedic Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Each participant data will be grouped for each cohort and averaged, so individual participant data is not necessary to perform a data analysis of the study.

REFERENCES:
- [Derived] Nguyen T, Hung VT, Hancock JU, Bailey D, Hess AV, Doarn M. Evaluating Patient Compliance With Woodcast and Thermoplast Splints After Thumb Carpometacarpal Arthroplasty: A Randomized Controlled Trial. Hand (N Y). 2026 Feb 8:15589447251415394. doi: 10.1177/15589447251415394. Online ahead of print. PMID 41656908